CLINICAL TRIAL: NCT03182634
Title: A Multiple Parallel Cohort, Multi-centre Phase IIa Trial Aiming to Provide Proof of Principle Efficacy for Designated Targeted Therapies in Patients With Advanced Breast Cancer Where the Targetable Mutation is Identified Through ctDNA
Brief Title: The UK Plasma Based Molecular Profiling of Advanced Breast Cancer to Inform Therapeutic CHoices (plasmaMATCH) Trial
Acronym: plasmaMATCH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ICR-CTSU/2015/10056
Record Dates: First submitted 2017-01-10; First posted 2017-06-09 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Fulvestrant; neratinib; capivasertib; olaparib; ceralasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort A - Extended-dose fulvestrant (Experimental): Fulvestrant 500mg IM on Cycle 1 Days 1, 8 and 15 and Cycle 2 onwards Days 1 and 15
  Interventions: Drug: Fulvestrant
- Cohort B - Neratinib (Experimental): Neratinib 240mg PO on a continuous schedule starting on Cycle 1 Day 1 AND in ER positive breast cancer, fulvestrant 500mg IM on Cycle 1 Days 1 and 15 and Cycle 2 onwards Day 1
  Interventions: Drug: Fulvestrant; Drug: Neratinib
- Cohort C - AZD5363 and fulvestrant (Experimental): AZD5363 400mg PO BID on a 7 day schedule of 4 days on treatment followed by 3 days off treatment AND fulvestrant 500mg IM Cycle 1 Days 1 and 15 and Cycle 2 onwards Day 1
  Interventions: Drug: Fulvestrant; Drug: AZD5363
- Cohort D - AZD5363 (Experimental): AZD5363 480mg PO BID on a 7 day schedule of 4 days on treatment followed by 3 days off treatment
  Interventions: Drug: AZD5363
- Cohort E - olaparib and AZD6738 (Experimental): AZD6738 160mg to be administered once daily on Days 1-7 of each cycle and olaparib 300mg to be administered twice daily on a continuous schedule starting on Cycle 1 Day 1.
  Interventions: Drug: Olaparib; Drug: AZD6738

INTERVENTIONS:
Drug: Fulvestrant
  Arms: Cohort A - Extended-dose fulvestrant; Cohort B - Neratinib; Cohort C - AZD5363 and fulvestrant
Drug: Neratinib
  Arms: Cohort B - Neratinib
Drug: AZD5363
  Arms: Cohort C - AZD5363 and fulvestrant; Cohort D - AZD5363
Drug: Olaparib
  Arms: Cohort E - olaparib and AZD6738
Drug: AZD6738
  Arms: Cohort E - olaparib and AZD6738

SUMMARY:
plasmaMATCH is a multi-centre phase IIa umbrella trial platform consisting of a ctDNA screening component and a therapeutic component. plasmaMATCH aims to assess whether ctDNA screening can be used to detect patient subgroups who will be sensitive to targeted therapies, and will also assess the safety and activity of the targeted treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Female.
2. Aged ≥ 18 years old.
3. Histologically confirmed invasive breast carcinoma.
4. Metastatic or recurrent locally advanced breast cancer that is not suitable for treatment with radical or curative intent.
5. Demonstrated progression of disease by radiological assessment or by clinical assessment within the last 6 weeks.
6. Measurable disease by RECIST v1.1.
7. Patients must have completed at least one prior line of treatment for advanced breast cancer and/or relapse within 12 months of completing (neo)adjuvant chemotherapy. Patients with HER2 positive breast cancer must have been treated with at least two courses of HER2 targeted therapy in the advanced setting (or one course if no further courses of HER2 targeted therapy are available locally).
8. Patient must either be suitable for a baseline biopsy of recurrent disease or have an archival biopsy of recurrent disease available. Patients are requested to consent to a baseline biopsy but if deemed unsafe by the Investigator, an archival biopsy of recurrent disease can be used instead. If it is deemed unsafe to proceed with baseline biopsy, and no archival recurrent disease biopsy is available, the patient will not be eligible for entry into the treatment cohort.
9. ECOG performance status ≤ 2.
10. Life expectancy >3 months in Cohorts A-D, >16 weeks in Cohort E.
11. Patients must be a) surgically sterile; b) have a sterilised sole partner; c) be postmenopausal; d) must agree to practice true abstinence; or e) must agree to use effective contraception during the period of trial treatment and be willing to do so for 6 months following the end of trial treatment. Effective contraception is defined as double barrier contraception (e.g. condom plus spermicide in combination with a diaphragm, cervical cap or intrauterine device). Ovarian suppression with an LHRH agonist is not a method of contraception.
12. Patients of childbearing potential should have a negative serum pregnancy test within 14 days prior to initiation of trial treatment.
13. At least 4 weeks washout period after the end of trial treatment on a different cohort within plasmaMATCH.
14. Adequate haematological, renal and hepatic function as defined by cohort-specific criteria in protocol.
15. For patients with ER positive breast cancer in Cohorts A, B and C: EITHER postmenopausal, as defined by at least one of the following criteria: Age >60 years; Age <60 years and cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and serum estradiol and follicle stimulating hormone (FSH) level within the laboratory's reference range for postmenopausal females; Documented bilateral oophorectomy; medically confirmed ovarian failure. OR Pre-/peri-menopausal (i.e. not meeting the criteria for being postmenopausal) if being treated with an LHRH agonist that was commenced at least 4 weeks prior to Cycle 1 Day 1, and continues on the LHRH agonist throughout the trial period.

NB. Additional eligibility criteria apply for entry into each treatment cohort.

Exclusion Criteria:

1. Prior treatment with radiotherapy (except for palliative reasons), endocrine therapy, immunotherapy, chemotherapy or IMPs during the previous 4 weeks (6 weeks for nitrosoureas, Mitomycin-C) before trial treatment, except for hormonal therapy with LHRH analogues, which are permitted, and bisphosphonates or RANK ligand antibodies that are permitted for the management of bone metastases.
2. Uncontrolled CNS disease (brain metastases or leptomeningeal disease). Patients with prior diagnosis of CNS metastases must be stable by clinical assessment having ceased steroids after prior treatment.
3. History of clinically significant or uncontrolled cardiac disease, including congestive heart failure, angina, myocardial infarction within the last 6 months or ventricular arrhythmia. Patients with a history of any of the above listed cardiac conditions judged not to be clinically significant by the local investigator must be notified to the trial team at the ICR-CTSU for approval by the CI and/or Cohort Lead.
4. Ongoing toxic manifestations of previous treatments Grade ≥1. Exceptions to this are alopecia or toxicities which in the opinion of the Investigator should not exclude the patient. Such cases should be clearly documented in the patient's notes by the Investigator.
5. Major surgery (excluding minor procedures, e.g. placement of vascular access) within 4 weeks of the first dose of trial treatment.
6. Pregnant or breastfeeding.
7. Any condition that according to the treating physician may compromise the patient's safety or the conduct of the trial.
8. Current malignancies of other types, with the exception of adequately treated in situ carcinoma of the cervix and basal or squamous cell carcinoma of the skin. Cancer survivors, who have undergone potentially curative therapy for a prior malignancy and have no evidence of the disease for 3 years or more are eligible for the trial.

NB. Additional eligibility criteria apply for entry into each treatment cohort.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1150 (Estimated)
Dates: Start 2016-12-15 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint for Cohorts A to E is confirmed objective response rate as defined by RECIST v1.1 for each cohort separately | up to 24 weeks

SECONDARY OUTCOMES:
Clinical benefit rate | up to 24 weeks
  A patient will be defined as having clinical benefit if they have either a complete/partial response or stable disease as defined by RECIST v1.1 lasting at least 24 weeks.
Progression free survival | up to 24 weeks
  PFS will be measured from the date of entry into the treatment cohort until first date of either confirmed progressive disease according to RECIST criteria or death.
Incidence of treatment-emergent adverse events (safety and tolerability) | through study completion, estimated average 1 year
  Incidence of treatment-emergent adverse events (safety and tolerability) will be assessed throughout the treatment period using the NCI CTCAE v4.0 and summarised in tabular format. Reported toxicities will be coded using MedDRA (current version). For each agent,the proportion of patients reporting a dose reduction/delay during trial treatment will be presented
Duration of response for each cohort | through study completion, estimated average 1 year
  The duration of response is measured from the time of first documentation of RECIST complete/partial response (whichever status is recorded first) until the first date that recurrence or progressive disease is objectively documented, taking as reference for progressive disease the smallest measurements recorded since the treatment started. Median duration of response and interquartile range will be presented along with its 95% confidence interval.
Frequency of mutations identified in ctDNA screening | Baseline
  The proportion of patients undergoing ctDNA screening who have each targetable mutation of interest will be presented.
The proportion of patients with a targetable mutation who enter a therapeutic component | Baseline
  The proportion of patients with a targetable mutation who enter the relevant therapeutic cohort will also be presented.
Agreement between ctDNA mutation status and tissue mutation status for patients entering the therapeutic component | Baseline
  The proportion of cancers with a ctDNA detected mutation that have a matching mutation on subsequent tissue biopsy will be presented with associated exact two-sided 95% confidence interval.
Maximum Plasma Concentration (Cmax) | Monthly up to 4 months
  Changes in Maximum Plasma Concentration during the treatment period for Cohorts A and B will be displayed graphically per patient. Values at specific time points will be summarised across all patients using the mean, standard deviation and range. Analyses will be performed separately for patients in Cohorts A and B.
Area Under the Curve (AUC) | Monthly up to 4 months
  Changes in area under the plasma concentration vs time curve during the treatment period for Cohorts A and B will be displayed graphically per patient. Values at specific time points will be summarised across all patients using the mean, standard deviation and range. Analyses will be performed separately for patients in Cohorts A and B.

CONTACTS AND LOCATIONS:
Locations (19):
- United Kingdom (19):
  - Royal Marsden Hosital, Sutton, England
  - Royal Bournemouth Hospital, Bournemouth
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Western General Hospital, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Clatterbridge Cancer Centre, Liverpool
  - Barts Health Trust, London
  - Royal Marsden Hospital, London
  - University College Hospital London, London
  - Kent Oncology Centre, Maidstone
  - Christie Hospital, Manchester
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Weston Park Hospital, Sheffield
  - University Hospitals Southampton NHS Foundation Trust, Southampton
  - Royal Cornwall Hospital, Truro

REFERENCES:
- [Derived] Kingston B, Cutts RJ, Bye H, Beaney M, Walsh-Crestani G, Hrebien S, Swift C, Kilburn LS, Kernaghan S, Moretti L, Wilkinson K, Wardley AM, Macpherson IR, Baird RD, Roylance R, Reis-Filho JS, Hubank M, Faull I, Banks KC, Lanman RB, Garcia-Murillas I, Bliss JM, Ring A, Turner NC. Genomic profile of advanced breast cancer in circulating tumour DNA. Nat Commun. 2021 Apr 23;12(1):2423. doi: 10.1038/s41467-021-22605-2. PMID 33893289
- [Derived] Turner NC, Kingston B, Kilburn LS, Kernaghan S, Wardley AM, Macpherson IR, Baird RD, Roylance R, Stephens P, Oikonomidou O, Braybrooke JP, Tuthill M, Abraham J, Winter MC, Bye H, Hubank M, Gevensleben H, Cutts R, Snowdon C, Rea D, Cameron D, Shaaban A, Randle K, Martin S, Wilkinson K, Moretti L, Bliss JM, Ring A. Circulating tumour DNA analysis to direct therapy in advanced breast cancer (plasmaMATCH): a multicentre, multicohort, phase 2a, platform trial. Lancet Oncol. 2020 Oct;21(10):1296-1308. doi: 10.1016/S1470-2045(20)30444-7. Epub 2020 Sep 10. PMID 32919527